CLINICAL TRIAL: NCT04870463
Title: Apical External Root Resorption Secondary to Orthodontic Forces and Individual Radicular Stress: Randomised Clinical Trial
Brief Title: Apical External Root Resorption Secondary to Orthodontic Forces and Individual Radicular Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Estrella1*
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Apical Root Resorption

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial of two parallel arms, that analysed the possible superiority of one treatment compared to the gold standard of reference
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gold Standard Group (Active Comparator): Patients treated with multi-braces fixed appliances and a conventional sequence of aligning and levelling arches (Ni-Ti arches with the same force in all sections)
  Interventions: Procedure: Maxillary and mandibular Cone Beam Computed Tomography record
- Intervention Group (Experimental): Patients treated with multi-braces fixed appliances and a different sequence of aligning and levelling arches (some arches provide individual forces for each group of teeth (incisors, premolars and molars))
  Interventions: Procedure: Maxillary and mandibular Cone Beam Computed Tomography record

INTERVENTIONS:
Procedure: Maxillary and mandibular Cone Beam Computed Tomography record — A Cone Beam Computed Tomography image of each patient of each group at three different moments of the study (baseline/T0, 8-9 months of treatment/T1 and end of treatment/T2)

SUMMARY:
The goal of this prospective clinical trial is to evaluate the possible superiority of a treatment compared to the gold standard of reference in Orthodontics.

DETAILED DESCRIPTION:
Apical external root resorption is defined as the loss of dental hard tissues such as dentine, cement and alveolar bone. This is considered an irrevocable effect associated to different factors, among which dental movement during orthodontic treatment is related.

This study suggest to compare root resorption after the use of two different types of alignment and levelling arches in orthodontics. Consecutive patients randomly chosen will be analysed after going through one of the two arches sequences:

1. Gold standard group: using arches that provide the same amount of force in all sections . 3M United® nickel-titanium arches (0.012, 0.014, 0.016 x 0.016, 0.020 x 0.020, 0.018 x 0.025 y 0.019 x 0.025)
2. Intervention group: using some arches that provide individual sectional forces for each dental group (incisors, premolars and molars). 3M United® nickel-titanium 0.012 and 0.014 arches and BioForce PLUS® arches (0.016 x 0.016, 0.020 x 0.020, 0.018 x 0.025 y 0.019 x 0.025).

All patients will be treated with multi-braces fixed appliances (0.022" technique and VictoryTM brackets).

Root resorption will be compared through CBCT (Cone Beam Computed Tomography) images made before the beginning of treatment (T0), after 8-9 months of the beginning of treatment (T1) and at the end of treatment (T2). Root resorption will be measured by the root volume and surface root morphology in each of the times scheduled.

ELIGIBILITY:
Study Population: patients undergoing orthodontic treatment in Orthodontic Department at Dental School of Universidad Complutense de Madrid.

Inclusion Criteria:

1. Completed permanent dentition (third molars are excluded)
2. Completed root formation
3. Need of orthodontic treatment

Exclusion Criteria:

1. Tooth agenesis in the anterior region (incisors)
2. Included or ankylosed teeth in the anterior region (incisors)
3. Periodontal pocket >3 mm in any anterior teeth (incisors)
4. Need of a combined surgical and orthodontic treatment
5. Root resorptions observed at the initial CBCT (in more than 3 teeth)
6. Delay of the treatment due to a external reason or complication during treatment
7. Systemic disease or cranio-facial malformation
8. Tooth fracture or restoration in the anterior region (incisors) at the beginning of treatment
9. Problems from roots such as lacerated root, trauma or fractures during treatment 10 Severe occlusal attrition

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Difference of volume of the apical portion of the root | Baseline/beginning treatment (T0), 34 weeks after beginning treatment (T1) and through treatment completion (T2)
  Measure of the 5 more apical mm3 of the root at each moment of treatment (T0, T1 and T2)

SECONDARY OUTCOMES:
Root volumen | Baseline/beginning treatment (T0), 34 weeks after beginning treatment (T1) and through treatment completion (T2)
  Measure of the total volume of each root at momento of treatment (T0, T1 and T2)
Root surface area | Baseline/beginning treatment (T0), 34 weeks after beginning treatment (T1) and through treatment completion (T2)
  Measure of the outer surface of the root dentine at momento of treatment (T0, T1 and T2)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Iglesias Linares, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Facultad de Odontología de la Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No